CLINICAL TRIAL: NCT06194734
Title: A Randomized, Controlled, Open-label, Multicenter Phase III Study to Evaluate the Efficacy and Safety of KC1036 Versus Investigator's Choice of Chemotherapy as Third-line Therapy in Patients With Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Study of KC1036 Versus Investigator's Choice of Chemotherapy in Patients With Advanced Esophageal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Konruns Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC1036-III-01
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Irinotecan; Docetaxel; S 1 (combination)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KC1036 (Experimental): KC1036 will be administrated.
  Interventions: Drug: KC1036
- Investigator's choice of chemotherapy (Active Comparator): Irinotecan, Docetaxel or S-1 will be administrated.
  Interventions: Drug: Irinotecan; Drug: Docetaxel; Drug: S-1

INTERVENTIONS:
Drug: KC1036 — KC1036 60mg QD orally, before a meal, continuous administration, 21 days as a cycle
  Arms: KC1036
Drug: Irinotecan — Irinotecan intravenously administered at 130-150 mg/m2 once every 2 weeks
  Arms: Investigator's choice of chemotherapy
Drug: Docetaxel — Docetaxel intravenously administered at 60-75 mg/m2 once every 3 weeks；
  Arms: Investigator's choice of chemotherapy
Drug: S-1 — S-1 orally administered 40-60mg Bid on Day 1 to Day 14 of every 3 weeks, 21 days as a cycle
  Other Names: Tegafur-gimeracil-oteracil potassium
  Arms: Investigator's choice of chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KC1036 versus investigator's choice of chemotherapy in patients with advanced recurrent or metastatic esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter phase III trial. Patients with advanced recurrent or metastatic esophageal squamous cell carcinoma that has received PD-1 or PD-L1 inhibitors and at least second-line systemic therapy will be randomized at a 1: 1 ratio to receive KC1036 or the investigator's choice of chemotherapy (Irinotecan/Docetaxel/S-1) until confirmed disease progression assessed by the RECIST V1.1 standard, death, intolerable toxicity, initiation of a new anti-tumor therapy, other reasons leading to treatment discontinuation as specified by protocol.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 to 75 years;
* Histologically or cytologically confirmed esophageal or esophageal-gastric junction squamous cell carcinoma;
* Patient with advanced recurrent or metastatic esophageal squamous cell carcinoma previously treated with a PD-1 or PD-L1 inhibitor and at least second-line systemic therapy;
* At least one measurable tumor lesion according to RECIST 1.1;
* Eastern Cooperative Oncology Group performance status score of 0 or 1;
* Life expectancy > 12 weeks;
* BMI≥16.0 and weight≥40 kg ;
* Adequate bone marrow, renal, and hepatic function;
* Female patients of childbearing potential with a negative blood pregnancy test completed within 7 days before randomization；
* Patients should participate in the study voluntarily and sign informed consent.

Exclusion Criteria:

* Any patient who is known to have untreated central nervous system (CNS) metastasis;
* Other kinds of malignancies within 5 years;
* Gastrointestinal abnormalities;
* Cardiovascular and cerebrovascular diseases;
* Prior therapies with vascular targeting inhibitor；
* Previously treated with Irinotecan, Docetaxel and Tegafur Gimeracil Oteracil Potassium；
* Involved in other clinical trials within 4 weeks before enrollment；Prior anti-tumor therapies with radiotherapy, immunotherapy, operation within 4 weeks before enrollment;Prior anti-tumor therapies with small molecule targeting drugs within 2weeks or 5 half-lives (whichever is longer) before enrollment; Prior anti-tumor therapies with chemotherapy within 3 weeks or 5 half-lives (whichever is longer) before enrollment;
* Presence of unresolved toxicities from prior anti-tumor therapy, defined as having not resolved to NCI CTCAE 5.0 Grade 0 or 1;
* Uncontrolled massive ascites, pleural or pericardial effusion;
* Severe infection within 4 weeks prior to randomization (CTCAE > Grade 2);
* Known history of human immunodeficiency virus (HIV) infection or current active hepatitis B or C infection;
* Pregnant or lactating women;
* Female subjects of child-bearing potential and male subjects of reproductive capacity who do not agree to use contraceptive measures during the study and for 6 months after the end of the study.
* Other patients are not eligible for enrollment assessed by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Baseline to study completion (approximately 24 months)
  OS is defined as the time from the start of randomization to death of any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (approximately 24 months)
  ORR is defined as the proportions of patients with a complete response (CR) or partial response (PR) according to RECIST 1.1.
Disease Control Rate (DCR) | Baseline to study completion (approximately 24 months)
  DCR is defined as the percentage of participants with a best overall complete response (CR), partial response (PR), or stable disease (SD) according to RECIST 1.1.
Duration of Response (DOR) | Baseline to study completion (approximately 24 months)
  DOR is defined as the time from first documented objective response (complete response (CR)or partial response (PR)) to the date of first documented disease progression (PD) or death.
Progression-free survival (PFS) | Baseline to study completion (approximately 24 months)
  PFS is defined as the time from the start of randomization to the date of the first documented progressive disease (PD) according to RECIST 1.1 or death.
Incidence of Adverse events (AEs) | Baseline to 30 days after the last dose of study treatment
  Assessed by treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) during the treatment assessed by NCI CTCAE 5.0.
Quality of Life (QOL) scores | Baseline to study completion (approximately 24 months)
  Quality of Life is a concept of comprehensive evaluation of the advantages and disadvantages of life. It mainly refers to the assessment of individual physiological, psychological and social functions, which is an important indicator of the effectiveness of medical and health care services.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, China